CLINICAL TRIAL: NCT02119169
Title: Pigtail Catheter: a Less Invasive Option for Pleural Drainage of Recurrent Hepatic Hydrothorax
Acronym: HH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, doctor, Tanta University
Organization: Tanta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mohamed Sharaf-Eldin; Tanta university hospital (Other Grant/Funding Number: tanta university hospital)
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pigtail catheter (Experimental): Pigtail catheter for pleural drainage of recurrent hepatic hydrothorax
  Interventions: Device: Pigtail catheter

INTERVENTIONS:
Device: Pigtail catheter — pigtail catheter for pleural drainage

SUMMARY:
The effectiveness of pigtail catheter as a less invasive option for pleural drainage in patients with resistant hepatic hydrothorax.

DETAILED DESCRIPTION:
Hepatic hydrothorax (HH) is defined as a transudative pleural effusion in patients with liver cirrhosis in the absence of cardiopulmonary disease. The estimated prevalence among patients with liver cirrhosis is approximately 5-6% (Baikati et al., 2014).

HH is an infrequent but a well-known complication of portal hypertension. Trans-diaphragmatic passage of ascitic fluid from peritoneal to the pleural cavity through numerous diaphragmatic defects has been shown to be the predominant mechanism in the formation of HH (Kumar&Kumar, 2014).

Patients with hepatic hydrothoraces often have few options (Goto et al., 2011). Diuretic-resistant HH could be managed with liver transplantation, transjugular intrahepatic portosystemic shunt (TIPS) or indwelling pleural catheters. However, tube thoracotomy and pleurodesis failed in most patients (Singh et al., 2013).

Case reports and small case series have reported a high rate of complications associated with chest tube placement for hepatic hydrothorax. The most common reported complications were acute kidney injury, pneumothorax, and empyema. Death has been recorded in some cases. Chest tube insertion for hepatic hydrothorax carries significant morbidity and mortality, with questionable benefit (Orman&Lok, 2009).

Pigtail catheter insertion is an effective and safe method of draining pleural fluid. Its use is safe and recommended for all cases of pleural effusion requiring chest drain except for empyema and other loculated effusions that yielded low success rate (Bediwy and Amer, 2012).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhotic liver and recurrent pleural effusion.
* Pleural fluid should be transudate according to Light's criteria:

  * Pleural fluid-to-serum protein ratio less than 0.5
  * Pleural fluid lactic dehydrogenase (LDH) less than 200 IU
  * Pleural fluid-to-serum LDH ratio and pleural fluid-to-high normal serum LDH ratio less than 0.6

Exclusion Criteria:

* Diagnosis of hepatocellular carcinoma or other neoplasm able to shorten life expectancy.
* Congestive heart failure.
* Recent (i.e. within the previous 2 weeks) episode of digestive hemorrhage.
* Exudative pleural effusion.
* Ascitic fluid or pleural fluid infection
* Platelet count below 50,000
* Prothrombin activity below 50%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in chest radiography | baseline, daily after treatment within admission

SECONDARY OUTCOMES:
Chest X-ray and any complications recorded | weekly in first month and monthly for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Sharaf-Eldin, professor, Principal Investigator — TUH; Adel S Bediwy, Professor, Study Director — TUH; Sherief M Abd-Elsalam, Doctor, Study Chair — TUH; Abdelrahman a kobtan, doctor, Study Chair — TUH
Locations (1):
- Tanta university hospital, Tanta, Egypt

REFERENCES:
- [Derived] Sharaf-Eldin M, Bediwy AS, Kobtan A, Abd-Elsalam S, El-Kalla F, Mansour L, Elkhalawany W, Elhendawy M, Soliman S. Pigtail Catheter: A Less Invasive Option for Pleural Drainage in Egyptian Patients with Recurrent Hepatic Hydrothorax. Gastroenterol Res Pract. 2016;2016:4013052. doi: 10.1155/2016/4013052. Epub 2016 Jun 2. PMID 27340399